CLINICAL TRIAL: NCT01994265
Title: Randomized Clinical Trial for the Prevention of Cognitive Impairment in Atrial Fibrillation Patients Treated With Dabigatran or Warfarin
Brief Title: Cognitive Impairment Related to Atrial Fibrillation Prevention Trial
Acronym: GIRAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Federal University of Minas Gerais (Other); Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Bruno Caramelli, Associate Professor of Cardiology, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USP/UFMG 2013
Record Dates: First submitted 2013-11-09; First posted 2013-11-25 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Cognition; Cognitive impairment; Anticoagulation; Dabigatran; Warfarin; Efficacy
MeSH Terms: conditions — Atrial Fibrillation; Cognitive Dysfunction | interventions — Warfarin; Dabigatran

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Warfarin (Active Comparator): Treatment with Warfarin once daily, taken at fast, to maintain INR between 2 and 3.
  Interventions: Drug: Warfarin
- Dabigatran (Active Comparator): Dabigatran 150 mg twice daily
  Interventions: Drug: Dabigatran

INTERVENTIONS:
Drug: Warfarin — Warfarin once daily, at fast, targeting INR between 2 and 3
  Other Names: Marevan, Coumadin
  Arms: Warfarin
Drug: Dabigatran
  Other Names: Dabigatran 150 mg twice daily
  Arms: Dabigatran

SUMMARY:
Cognitive and functional decline observed in atrial fibrillation (AF) patients are related to thrombotic and/or cardioembolic events. Use of warfarin for the prevention of stroke in AF patients, despite effective, remains beyond desired levels because of interactions with food and fluctuations in blood levels. Because of a more stable anticoagulation state, Dabigatran may offer better protection against thrombotic phenomenon and, consequently, mitigate the process of cognitive and functional compromise.

DETAILED DESCRIPTION:
This will be a prospective parallel study including two hundred atrial fibrillation patients > 65 years old and scoring CHADS2VASc > 1. Patients will be randomized to receive Warfarin (INR between 2 and 3) or Dabigatran (150 mg twice daily) for two years. After one year and at the end of the study, individuals will be evaluated regarding cognitive endpoints following the National Institute of Neurological Disorders and Stroke-Canadian Stroke Network Vascular Cognitive Impairment Harmonization Standards (Hachinski et al. Stroke 2006;37:2220-2241). The investigators will use the 60 minutes evaluation protocol complemented by the Montreal Cognitive Assessment (MoCA).

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation
* CHA2DS2-VASc Score for Atrial Fibrillation Stroke Risk (CHADS2VASc) greater than 1

Exclusion Criteria:

* Heart valve disease
* Previous Stroke or Transient ischemic attack
* Cognitive impairment or any severe neurological disorder
* Major surgery in the last 30 days
* Planned elective surgery in the next three months
* Intracranial, ocular, spinal, retroperitoneal, or articular bleeding without trauma.
* Gastrointestinal bleeding in the last 12 months
* Symptomatic gastric ulcer
* Hemorrhagic disease
* Use of thrombolytics
* Uncontrolled hypertension
* Active cancer
* Contraindication for Warfarin use
* Reversible causes of atrial fibrillation
* Creatinine clearance < 30 ml/min
* Active endocarditis
* Active hepatitis
* Severe anemia
* Left ventricle ejection fraction < 35%

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-11-07; Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Cognitive impairment | Two years
  Cognitive impairment at two years, independently of stroke or other cerebrovascular events.

SECONDARY OUTCOMES:
Number of Participants with less important alteration in coagulation test as a Measure of Safety | Two years
  Comparison of thrombin generation test between the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Caramelli, Professor, Principal Investigator — Heart Institute, University of Sao Paulo, Brazil
Locations (2):
- Brazil (2):
  - Federal Univeristy of Minas Gerais, Belo Horizonte, Minas Gerais
  - Heart Institute - University of São Paulo, São Paulo

REFERENCES:
- [Derived] Caramelli B, Yu PC, Cardozo FAM, Magalhaes IR, Spera RR, Amado DK, Escalante-Rojas MC, Gualandro DM, Calderaro D, Tavares CAM, Borges-Junior FA, Pastana AF, Matheus MG, Brucki SMD, Rodrigues ACO, Nitrini R, Caramelli P. Effects of dabigatran versus warfarin on 2-year cognitive outcomes in old patients with atrial fibrillation: results from the GIRAF randomized clinical trial. BMC Med. 2022 Oct 26;20(1):374. doi: 10.1186/s12916-022-02563-2. PMID 36284318